CLINICAL TRIAL: NCT04314622
Title: A Randomized, Double-Blind, Placebo-controlled Study of Supaglutide on the Safety, Pharmacokinetics and Pharmacodynamics, and Efficacy in Chinese Patients With Type 2 Diabetes.
Brief Title: A Study of Supaglutide in Chinese Type 2 Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Collaborators: Shanghai 6th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YN011B
Record Dates: First submitted 2020-03-11; First posted 2020-03-19 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supaglutide (Part A) (Experimental): Four investigational doses of Supaglutide administered weekly (or bi-weekly) and subcutaneously (SC) in T2DM patients.
  Interventions: Drug: Supaglutide
- Placebo(Part A) (Placebo Comparator): Placebo administered weekly (or bi-weekly) and SC in T2DM patients.
  Interventions: Drug: Placebo
- Supaglutide (Part B) (Experimental): Two investigational doses of Supaglutide administered weekly (or bi-weekly) and SC in T2DM patients.
  Interventions: Drug: Supaglutide
- Placebo (Part B) (Placebo Comparator): Placebo administered weekly (or bi-weekly) and SC in T2DM patients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Supaglutide — Administered SC
  Other Names: Diabegone
  Arms: Supaglutide (Part A); Supaglutide (Part B)
Drug: Placebo — Administered SC
  Arms: Placebo (Part B); Placebo(Part A)

SUMMARY:
A study on the safety, efficacy, pharmacokinetics and pharmacodynamics of Supaglutide dosing weekly and bi-weekly in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Have diagnosed with type 2 diabetes for at least 3 months before enrollment.
2. Have diet and exercise intervention only (for part A and part B) or been treated with stable dose of metformin as monotherapy for at least 3 months (for part B only)
3. Have HbA1c ≥7.0% and ≤10.0% as assessed by the central laboratory.
4. Have a body mass index (BMI) of 20-40 kilograms per square meter (kg/m^2).

Exclusion Criteria:

1. Type 1 diabetes (T1D).
2. Evidences of fasting C-peptide levels<0.81 ng/mL.
3. History of trauma, infection or surgery within a month;
4. History of blood donation, blood transfusion or losing more than 450 ml blood within 3 months.
5. History of the severe cardiovascular conditions, gastrointestinal diseases, blood system diseases, pancreatitis, or malignant tumors.
6. Evidence of abnormal thyroid function within 6 months before screening.
7. Positive test results in HBsAg, HCVAB, HIVAB or TPAB.
8. History of serious mental illness.
9. History of drug or alcohol abuse.
10. History of a transplanted organ, acquired or congenital immune system diseases.
11. Allergy to active ingredients or excipients of the test drug.
12. Evidence of abnormal result of laboratory examination according to the judgment of researchers.
13. Participated in any interventional medical, surgical, or pharmaceutical study within 3 months prior to entry into the study.
14. Previously completed or withdrawn from this study after providing informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline, 7 weeks, 17weeks
  Change from Baseline in Hemoglobin A1c (HbA1c)
Adverse Events | Baseline , through 12 weeks for part A; Baseline, through 17 weeks for part B
  Number of Adverse Events
Vital Sign | Baseline , through 12 weeks for part A; Baseline, through 17 weeks for part B
  Assessments of Vital Sign
Laboratory Tests | Baseline , through 12 weeks for part A; Baseline, through 17 weeks for part B
  Assessments of Laboratory Tests
12-lead ECGs | Baseline , through 12 weeks for part A; Baseline, through 17 weeks for part B
  Assessments of 12-lead ECGs
Immunogenicity Tests | Baseline , through 12 weeks for part A; Baseline, through 17 weeks for part B
  Assessments of Immunogenicity Tests

SECONDARY OUTCOMES:
HbA1c <7% | Baseline, 7 weeks, 17weeks
  Percentage of Participants Achieving HbA1c Target <7.0%
Glycosylated Albumin | Baseline, 7 weeks, 17weeks
  Changes from Baseline in Glycosylated Albumin
Fasting Blood Glucose | Baseline, 7 weeks, 17weeks
  Changes from Baseline in Fasting Blood Glucose
Fasting Blood Insulin | Baseline, 7 weeks, 17weeks
  Changes from Baseline in Fasting Blood Insulin
Fasting Blood C-peptide | Baseline, 7 weeks, 17weeks
  Changes from Baseline in Fasting Blood C-peptide
Blood Lipid | Baseline, 7 weeks, 17weeks
  Changes from Baseline in Blood Lipid
Body Weight | Baseline, 7 weeks, 17weeks
  Changes from Baseline in Body Weight
Pharmacokinetics (PK): Area Under the Curve | Day1, Day8, Day36 and Day43: Predose, 3, 6, 12, 24, 48, 72, 96, 168 and 336 hours post dose (in part A)
  Area Under the Plasma Drug Concentration-Time Curve from Zero to Infinity (AUC0-∞)
Pharmacokinetics (PK): t½ of Supaglutide | Day1, Day8, Day36 and Day43: Predose, 3, 6, 12, 24, 48, 72, 96, 168 and 336 hours post dose (in part A)
  Terminal Elimination Half-life in Plasma (t½)
PK: Tmax of Supaglutide | Day1, Day8, Day36 and Day43: Predose, 3, 6, 12, 24, 48, 72, 96, 168, and 336 hours post dose (in part A)
  Time to Maximum Plasma Concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, Doctor, Principal Investigator — Department of Endocrinology and Metabolism, Shanghai Sixth People's Hospital; Yuqian Bao, Doctor, Principal Investigator — Department of Endocrinology and Metabolism, Shanghai Sixth People's Hospital
Locations (1):
- The Affiliated Zhongda Hospital of Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lou YR, Xu YL, Xiong Y, Deng C, Wang Q. Population Pharmacokinetics of Efsubaglutide Alfa in Healthy Subjects and Subjects with Type 2 Diabetes. Clin Pharmacokinet. 2025 Apr;64(4):533-552. doi: 10.1007/s40262-025-01475-7. Epub 2025 Feb 17. PMID 39961992